CLINICAL TRIAL: NCT02718274
Title: HIV Self-testing Africa (STAR) Malawi: General Population - A Cluster Randomized Trial of Providing HIV and Self-testing Kits Through Community-based Distribution Agents
Brief Title: HIV Self-Testing Africa (STAR) Malawi: General Population
Acronym: STAR Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: UNITAID (Other); Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other); Liverpool School of Tropical Medicine (Other); University College, London (Other); Population Services International (Other); World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10566
Record Dates: First submitted 2016-03-18; First posted 2016-03-24 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2017-08

CONDITIONS: HIV
Keywords: HIV self-testing; Malawi; HIV
MeSH Terms: interventions — Drug Packaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Standard of care.
- Self-testing (Active Comparator): Community-Based Distribution Agents (CBDAs) in the HIV Self-Testing (HIVST) Arm villages will be trained to provide HIVST services as well as reproductive health services.
  Interventions: Device: OraQuick ADVANCE HIV I/II test kits, packaged for self-use (manufactured in Thailand)
- Self-testing + home HIV care home initiation (Active Comparator): CBDAs will be trained to provide HIV Self-Testing plus offer home assessment and HIV care initiation (first assessment and first 14 days of HIV care medications), with this additional intervention aimed at facilitating linkage into care.
  Interventions: Device: OraQuick ADVANCE HIV I/II test kits, packaged for self-use (manufactured in Thailand); Other: Home-based initiation of ARVs

INTERVENTIONS:
Device: OraQuick ADVANCE HIV I/II test kits, packaged for self-use (manufactured in Thailand) — Community based distribution of self-tests
  Arms: Self-testing; Self-testing + home HIV care home initiation
Other: Home-based initiation of ARVs — Home-based initiation of ARVs by study nurse linked to follow-up at clinic
  Arms: Self-testing + home HIV care home initiation

SUMMARY:
The aim of this project is to investigate the feasibility, affordability as well as the health and social impact of introducing HIV self-testing to rural communities through existing community-based volunteer services.

DETAILED DESCRIPTION:
The aim of this project is to investigate the incremental costs and health benefits of adding HIVST to the remit of existing cadres of community volunteers in the general population in Malawi.

Specific objectives are to:

1. Validate the use of the OraQuick HIVST product in rural settings, establish preferences and social harms reporting systems, and conduct baseline surveys.
2. Carry out a pragmatic cluster-randomised trial with ART clinics and their catchment populations, including CBDAs, as the unit of randomisation.
3. Evaluate the impact of adding HIVST into the remit of VMMC mobilisers on demand for VMMC
4. Establish the expected costs and benefits of introducing HIVST to Malawi through economic and mathematical modelling.
5. Conduct interviews with policy-makers to prepare for national scale-up of HIVST and support the market introduction of quality-assured HIVST products.

CRCT METHODOLOGY/STUDY DESIGN

First stage randomization: HIVST v. SOC. The main study will be a cluster-randomised trial in up to 5 high HIV prevalence districts (provisionally Blantyre, Machinga, Mwanza, Neno and Thyolo) that already have community-based reproductive health services provided by PSI under funding provided by the German Technical Cooperation Agency (GTZ). This programme supports volunteers to socially-market reproductive and child health products in villages, with products stored and managed by collaborating primary care clinics. The unit of randomisation is the Primary Care + ART Clinic and surrounding catchment area villages to clinic. CBDAs in the HIVST Arm villages will be trained to provide HIVST services as well as reproductive health services. CBDAs in the SOC Arm villages will remain with reproductive health services only. Two separate units of evaluation will be pre-defined before randomisation: one or two evaluation villages that will have baseline-final household surveys, and a wider catchment area including all villages with CBDA activities.

Second stage randomization: HIVST with and without home assessment. Villages in the HIVST intervention area will be randomised to either HIVST only, or to HIVST plus offer of home assessment and HIV care initiation (first assessment and first 14 days of HIV care medications) with this additional intervention aimed at facilitating linkage into care.

CRCT SAMPLE SIZE

This trial has one primary and one secondary outcome, with a number of other analyses to be specified in the Statistical Analysis Plan. The sample size considerations here relate to the main Primary Outcome (comparison between arms of recent HIV testing).

A survey sample of 250 to 500 adults per cluster will provide sufficient power for a two sample comparison of unmatched proportions for HTC coverage was performed across the intervention and control arms to determine the number of clusters per arm.

The cluster size is based on the typical size of a rural village (250-500 people) from previous experience in Malawi. Using 2010 DHS data, baseline rates for individuals tested in the last 12 months is estimated at 25% to 40%, with a 45% to 60% predicted effect size in the intervention arm compared to the control arm. Baseline coverage for individuals who have ever tested is estimated at 42% to 60% with predicted effect size 30%-45%.

Figures 10 and 11 in the full protocol contain a table of scenarios for each of the outlined assumptions. To detect a 50% increase in rate of people testing in the past 12 months and a 45% increase in the percentage of people who have ever tested in the intervention villages, there should be approximately 8 clusters per arm and approximately 4,000 participants total. This study will aim to reach 10 clusters per arm and 5,000 participants to provide contingency for a lower than anticipated effect size.

FORMATIVE RESEARCH

Formative research will be conducted before the beginning of the cRCT, including (1) cognitive interviews to assess the suitability existing IFUs in this population and modify IFUs as needed; (2) key informant interviews to help identify needs of stakeholders working in this area; (3) community mapping to identify local services.

Cognitive interviewing to validate IFUS. Convenience sampling will be used to recruit clients from VCT clinics for the cognitive interviews. Eligibility criteria include clients who are 16 years or older, and willing to provide written informed consent for participation in the study. A witnessed thumbprint will be sufficient for those who are unable to read or write. Participants will be purposively selected to ensure a range in location and literacy level. Four to 12 participants will be recruited for each iteration of the cognitive interviews, with a maximum of 12 iterations of adaptation and trial of the intended IFUs (n = 144). Cognitive interviewing and iterative adaptation will continue until saturation occurs and no further modifications to user materials are made.

Key informant interviews. We will conduct key informant interviews to inform our understanding of needs through key informant interviews with stakeholders working in HIV policy, product regulation and HIV implementation. Approximately 45 participants will be selected purposively through snowball sampling for the KIIs. MLW-LSHTM, using their professional networks and PSI country staff, will identify appropriate stakeholders. Interviews will be with written informed consent, will use semi-structured questionnaires and will be audiotaped.

Community mapping. Primary care clinics and evaluation villagers will be selected in consultation with the program lead for PSI's CBDA programme, and in consultation with the relevant District Health Offices, Primary care clinics and the CBDAs themselves.Once villages have been selected, preliminary mapping exercises will be initiated including demarcation of the village boundaries and location of dwellings with geographical position system (GPS) and a brief household-level questionnaire (name of household head, demographics of household members).

PILOT STUDY

Two villages not included in the main study will be selected from rural Blantyre or Thyolo for pilot studies of accuracy and acceptability. From these villages, 200 to 250 participants in total will be recruited from either randomly selected households (n = 150-200) or community peer groups (n = 48) for the accuracy and acceptability studies .Participants who opt to self-test as well as undergo standard HTC will be given a HIVST kit and a test results forms to record their own reading of the results. They will then be provided with a demonstration and instructions before carrying out the self-test procedure in a private room and completing the test results forms. Participants who themselves recognise that they have made a user error or find that their first result is uninterpretable will be given a second test kit to repeat the procedure if they wish to do so.

Following self-testing, trained HTC counsellors will record their own reading of the test kit before completing the standard HTC process (parallel Unigold and Determine finger prick blood) and entering the results of blood-based testing. All patients testing HIV+ve will be referred to HIV care services.

PILOT STUDY SAMPLE SIZE

For the pilot study, 150 to 200 adults will be recruited from a random selection of 60 to 80 households (with an estimated 2-5 adults per household) using randomly selected GPS waypoints. All household members aged 16 years or older will be asked for written consent to answer a brief questionnaire (socio demographics, past HIV testing experience, chronic care including ART) and will be offered HIVST followed immediately by confirmatory HTC. Parental consent will be taken for 16 and 17-year-olds and witnessed thumbprint for individuals unable to read or write.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or above
* Usual residence within a study PHC catchment area
* Able and willing to provide oral consent to HTC

Exclusion Criteria:

* Age 15 years or below
* Usual residence outside of the intervention cluster

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5504 (Actual)
Dates: Start 2016-04; Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Comparison between randomisation arms in coverage of recent (within the last 12 months) HIV testing among adult (16 years and above) village residents 12 months after the initiation of the intervention, measured by self-report through a household survey | 13 months
Comparison between randomisation arms of number of adult (16 yrs or older) village residents disclosing a positive results to the CBDA during months 1 to 12 of intervention, with a confidential post-test log book used to capture these data | 13 months

SECONDARY OUTCOMES:
Comparison between randomisation arms of ART initiation rates for adult (16 yrs or older) cluster residents, during months 1 to 12 of intervention, measured using clinic data extraction | 13 months
Comparison between randomisation arms of ART initiation rates for adult (16 yrs or older) village residents during months 1 to 12 of intervention, with ART clinic records used for this assessment | 13 months

CONTACTS AND LOCATIONS:
Locations (1):
- Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Indravudh PP, Fielding K, Chilongosi R, Nzawa R, Neuman M, Kumwenda MK, Nyirenda R, Johnson CC, Taegtmeyer M, Desmond N, Hatzold K, Corbett EL. Effect of door-to-door distribution of HIV self-testing kits on HIV testing and antiretroviral therapy initiation: a cluster randomised trial in Malawi. BMJ Glob Health. 2021 Jul;6(Suppl 4):e004269. doi: 10.1136/bmjgh-2020-004269. PMID 34275866
- [Derived] Johnson C, Kumwenda M, Meghji J, Choko AT, Phiri M, Hatzold K, Baggaley R, Taegtmeyer M, Terris-Prestholt F, Desmond N, Corbett EL. 'Too old to test?': A life course approach to HIV-related risk and self-testing among midlife-older adults in Malawi. BMC Public Health. 2021 Apr 3;21(1):650. doi: 10.1186/s12889-021-10573-7. PMID 33812381
- [Derived] Kumwenda MK, Johnson CC, Choko AT, Lora W, Sibande W, Sakala D, Indravudh P, Chilongosi R, Baggaley RC, Nyirenda R, Taegtmeyer M, Hatzold K, Desmond N, Corbett EL. Exploring social harms during distribution of HIV self-testing kits using mixed-methods approaches in Malawi. J Int AIDS Soc. 2019 Mar;22 Suppl 1(Suppl Suppl 1):e25251. doi: 10.1002/jia2.25251. PMID 30907508
- [Derived] Neuman M, Indravudh P, Chilongosi R, d'Elbee M, Desmond N, Fielding K, Hensen B, Johnson C, Mkandawire P, Mwinga A, Nalubamba M, Ncube G, Nyirenda L, Nyrienda R, Kampe EOI, Taegtmeyer M, Terris-Prestholt F, Weiss HA, Hatzold K, Ayles H, Corbett EL. The effectiveness and cost-effectiveness of community-based lay distribution of HIV self-tests in increasing uptake of HIV testing among adults in rural Malawi and rural and peri-urban Zambia: protocol for STAR (self-testing for Africa) cluster randomized evaluations. BMC Public Health. 2018 Nov 6;18(1):1234. doi: 10.1186/s12889-018-6120-3. PMID 30400959